CLINICAL TRIAL: NCT06140797
Title: Prehabilitation Combined With Enhanced Recovery After Surgery (PREERAS) in the Chinese Elderly With Spine Surgery
Brief Title: Pre-operative Risk Assessment Combined With Targeted Intervention in the Chinese Elderly With Spine Surgery
Acronym: PRACTICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: lushibao
Record Dates: First submitted 2023-11-08; First posted 2023-11-20 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Spine Degeneration; Spine Fusion; Frailty Syndrome
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PREERAS group (Experimental): Pre-operative risk assessment combined with targeted intervention During the planning phase of the study, we assembled a multidisciplinary team consisting of geriatrician, spine surgeons, nurses, rehabilitation specialists, anesthesiologists, neurologists, nutritionist, and social workers. Then, the multimodal prehabilitation combined with perioperative ERAS care (PREERAS) programme was conducted based on previous studies and surgical guideline.
  Participants randomised to the intervention group will receive PREERAS management. PREERAS mainly consists of geriatric assessment, Vivifrail multicomponent exercise, nutritional intervention, cognitive prehabilitation and brain protection.
  Interventions: Combination Product: Multimodal prehabilitation combined with perioperative ERAS care（PREERAS）
- Control group (No Intervention): The control group will receive standard of enhanced recovery after surgery (ERAS) care that is provided as part of the perioperative surgical procedure and subsequent rehabilitation

INTERVENTIONS:
Combination Product: Multimodal prehabilitation combined with perioperative ERAS care（PREERAS） — Pre-admission risk assessment and targeted intervention provided by multidisciplinary team
  Arms: PREERAS group

SUMMARY:
With the extended life expectancy of the Chinese population and improvements in surgery and anesthesia techniques, the number of aged patients undergoing surgery has been increasing annually. However, safety, effectiveness, and quality of life of aged patients undergoing surgery are facing major challenges. This prospective, multi-center, randomized, controlled study aims to construct a prehabilitation combined with enhanced recovery after surgery program which includes pre-operative risk assessment and targeted intervention.

DETAILED DESCRIPTION:
According to the United Nations 2022 Revision of World Population Prospects, the proportion of people over 65 years of age is expected to increase from approximately 9.7% in 2022 to 16.4% in 2050. The burden of spine disorders has increased substantially with the unprecedented aging population and the increase in life expectancy. Recent studies using multicenter data have showed that the increase in spinal fusions for spinal degenerative diseases was highest among patients over 75 years. Despite improved quality-adjusted life years and symptomatic benefits with spinal fusion surgery, there is an observed excess of adverse postoperative outcomes in older patients (aged 75 years and older) compared with younger patients. Enhanced Recovery After Surgery (ERAS) involves multidisciplinary perioperative measures to reduce surgical stress responses and improve perioperative outcomes and postoperative recovery. However, ERAS does not include preoperative comprehensive interventions to address or optimize the comorbidities, malnutrition, decreased functional capacity that are commonly present in older patients. In addition to the comorbid risk factors that older patients share with younger ones, older patients may also have malnutrition and cognitive or functional impairment. In older patients, the accumulation of geriatric frailty and various geriatric syndromes leads to decreased physiological reserves, resulting in a challenging recovery process after spine surgery. A possible way to overcome this variability and therefore to identify the patients at risk of adverse events (AEs) is to use specific tools developed by geriatricians and included in the so-called Comprehensive Geriatric Assessment (CGA).

CGA is a multi-dimensional diagnostic process designed to evaluate an elderly patient's medical, psychosocial, functional, and environmental resources and links them with an overall plan of treatment and follow-up. Guidelines and recommendations have addressed the importance of combined geriatric assessment and operational risks as an alternative to traditional preoperative assessment in elderly patients. The value of CGA in predicting long-term quality-of-life and functional decline has been demonstrated in previous studies on cancer surgery and hip fracture surgery; however, few studies on spine surgery included CGA in their analyses. Although some items in CGA, such as frailty and depression, have been shown to be associated with postoperative complications after spinal surgery, few studies have performed a complete evaluation of CGA in older patients. The reluctance of site leads and participants to use the comprehensive tool may reflect the volume of information it included, which may have made it difficult for clinicians to identify and use relevant sections. Most older people who have spinal disorders are frail, have comorbidities, and show a functional deterioration, which adversely affects quality of life and delays postoperative rehabilitation. Prehabilitation programs aim to strengthen patients physically and mentally before surgery by addressing modifiable risk factors during the preoperative period while they are waiting for surgery thereby filling this existing gap. Emerging evidence suggests a benefit of prehabilitation before major abdominal and cardiothoracic surgery. However, high-level evidence supporting the integration of CGA-based prehabilitation into ERAS program is still limited, particularly within the context of spine surgery.

The overall aim of this work is to examine the effect of multimodal prehabilitation combined with perioperative ERAS care (PREERAS) compared to only-ERAS in older patients (aged 75 years and older) scheduled for spinal fusion surgery. The study hypothesizes that the PRE-ERAS program will be more effective than only-ERAS care in improving postoperative clinical outcomes and patients-reported outcomes (PRO).

Study design and setting This study is a prospective, multicenter, parallel, randomized, controlled study. This study will be carried out in three tertiary teaching hospitals, including Xuanwu Hospital, Peking University First Hospital, and Beijing Friendship Hospital. The patients of control group will receive the established perioperative ERAS care. Pre-admission intervention include education on smoking and excessive drinking cessation, available counseling services, optimization of chronic disease, and nutritional assessment and support (only through nutritional education). Participants randomized to the intervention group will receive PREERAS management. PREERAS mainly consists of geriatric assessment, Vivifrail multicomponent exercise, nutritional intervention, cognitive prehabilitation and brain protection. The study will start in April 2024. The recruitment period will be 20 months, with a follow-up of 90 days. The results of the study will be expected in December 2025.

Primary outcomes: The primary outcome is the Comprehensive Complication Index (CCI; scores range from 0 to 100, with a score of 100 being death as a result of complications) which integrates all complications with their respective severities on a continuous scale ranging from 0 (no burden due to complications) to 100 (death as a result of complications). The CCI is based on the complication grading by the Clavien-Dindo Classification and captures every complication that occurred after an intervention. Postoperative complications were recorded to 90-day after surgery (definitions provided in supplementary table 1) and scored by severity using the Clavien-Dindo classification. The CCI was derived from these scores using the CCI calculator available online (http://www.assessurgery.com). Previous studies have validated the CCI as a measure of postoperative morbidity, suggesting that it offers a more comprehensive and sensitive endpoint for surgical research compared to traditional morbidity measures, such as the overall rate of complications or the rate of severe complications.

Secondary outcomes: Pain levels and pain-related function and activity limitation will be measured by visual analogue scale (VAS) and Oswestry/Neck disability index (ODI/NDI). Health- related quality of life will be evaluated by EuroQol Five Dimensions Questionnaire (EQ-5D, 0 = worst health and 100 = best health). Physical function will be assessed using 6 m walking speed and hand grip strength. Patient satisfaction will be measured using the North American Spine Society (NASS) satisfaction scale, measured on a scale of 1-4, with 1 indicating most satisfied and 4 indicating least satisfied. Answers on the satisfaction scale are as follows: The treatment met my expectations (score 1); I don't not improve as much as I had hoped, but I would undergo the same treatment for the same outcome (score 2); I don't improve as much as I had hoped, and I would not undergo the same treatment for the same outcome (score 3); I am the same or worse than before treatment (score 4). Data regarding primary and total length of hospital stay, non-home discharge, readmissions, and unplanned readmission within 90 days after surgery will be followed up. The discharge criteria for all patients were as follows: (1) preoperative symptoms are entirely or mainly relieved, or treatment has met the patient's expectations; (2) patients have no surgery-related complications, or the postoperative complications have been controlled, and (3) no further treatment is required.

ELIGIBILITY:
Inclusion Criteria:

1. patients who voluntarily sign the informed consent form; (2) elective spinal fusion surgery for degenerative spinal disorders; (3) no severe cognitive impairment (MoCA score ≥ 8).

   Exclusion Criteria:

   Patients (1) are scheduled to undergo emergency or day surgery,
2. have urgent condition that needs to be managed before the surgery,
3. are unable to cooperate with preoperative assessment,
4. have spinal fractures, metastasis, and spinal infections,
5. unable to understand or participate safely in intervention program,
6. participate in another study that may affect the study.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 164 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Comprehensive Complication Index | up to 90 days after surgery
  The Comprehensive Complication Index (CCI) is based on the complication grading by the Clavien-Dindo Classification and captures every complication that occurred after an intervention. Postoperative complications were recorded to 90-day after surgery (definitions provided in supplementary table 1) and scored by severity using the Clavien-Dindo classification. The CCI was derived from these scores using the CCI calculator available online (http://www.assessurgery.com). Previous studies have validated the CCI as a measure of postoperative morbidity, suggesting that it offers a more comprehensive and sensitive endpoint for surgical research compared to traditional morbidity measures, such as the overall rate of complications or the rate of severe complications.

SECONDARY OUTCOMES:
Neck/Oswestry disability index | up to 90 days after surgery
  Oswestry disability index (0 - 100 points, a higher total score reflects higher disability) for lumbar surgery and Neck disability index ( 0 - 100 points, a higher total score reflects higher disability] for cervical surgery).
EuroQol Five Dimensions Questionnaire (EQ-5D) | up to 90 days after surgery
  Health- related quality of life will be evaluated by EuroQol Five Dimensions Questionnaire (EQ-5D, 0 = worst health and 100 = best health).
6 m walking speed | up to 90 days after surgery
  Time in seconds to walk 6 m at usual pace expressed as m/s
North American Spine Society scores | up to 90 days after surgery
  Patient satisfaction will be measured using the North American Spine Society (NASS) satisfaction scale, measured on a scale of 1-4, with 1 indicating most satisfied and 4 indicating least satisfied. Answers on the satisfaction scale are as follows: The treatment met my expectations (score 1); I don't not improve as much as I had hoped, but I would undergo the same treatment for the same outcome (score 2); I don't improve as much as I had hoped, and I would not undergo the same treatment for the same outcome (score 3); I am the same or worse than before treatment (score 4).
Primary and total length of hospital stay | up to 90 days after surgery
  The discharge criteria for all patients are as follows: (1) preoperative symptoms are entirely or mainly relieved, or treatment has met the patient's expectations; (2) patients have no surgery-related complications, or the postoperative complications have been controlled, and (3) no further treatment is required.
Rates of non-home discharge | up to 90 days after surgery
  The non-home discharge includes inpatient rehabilitation, complex continuing care (CCC), long term care (LTC), and transferred to another inpatient setting.
Rates of unplanned readmission | up to 90 days after surgery
  90-days unplanned readmission for complications or pain
Hand grip strength | up to 90 days after surgery
  Grip strength will be measured in both hands. The patients sit in a comfortable position, with their elbows extended, and squeezed the dynamometer with maximum strength. The grip strength will be measured twice for both hands, with a short break in between. The best performance, regardless of hand dominance, will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Shibao Lu, Study Chair — Xuanwu Hospital, Beijing; Shuaikang Wang, Study Director — Capital Medical University; Chun-De Li, Principal Investigator — Peking University First Hospital; Yong Yang, Principal Investigator — Beijing Friendship Hospital
Locations (3):
- China (3):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kassebaum DG, Judkins MP, Griswold HE. Stress electrocardiography in the evaluation of surgical revascularization of the heart. Circulation. 1969 Sep;40(3):297-313. doi: 10.1161/01.cir.40.3.297. No abstract available. PMID 5810888
- [Background] Martin BI, Mirza SK, Spina N, Spiker WR, Lawrence B, Brodke DS. Trends in Lumbar Fusion Procedure Rates and Associated Hospital Costs for Degenerative Spinal Diseases in the United States, 2004 to 2015. Spine (Phila Pa 1976). 2019 Mar 1;44(5):369-376. doi: 10.1097/BRS.0000000000002822. PMID 30074971
- [Background] Rivier C, Shen GH. In the rat, endogenous nitric oxide modulates the response of the hypothalamic-pituitary-adrenal axis to interleukin-1 beta, vasopressin, and oxytocin. J Neurosci. 1994 Apr;14(4):1985-93. doi: 10.1523/JNEUROSCI.14-04-01985.1994. PMID 8158253
- [Background] Karsy M, Chan AK, Mummaneni PV, Virk MS, Bydon M, Glassman SD, Foley KT, Potts EA, Shaffrey CI, Shaffrey ME, Coric D, Asher AL, Knightly JJ, Park P, Fu KM, Slotkin JR, Haid RW, Wang M, Bisson EF. Outcomes and Complications With Age in Spondylolisthesis: An Evaluation of the Elderly From the Quality Outcomes Database. Spine (Phila Pa 1976). 2020 Jul 15;45(14):1000-1008. doi: 10.1097/BRS.0000000000003441. PMID 32097272
- [Background] Whittle AK, Kalsi T, Babic-Illman G, Wang Y, Fields P, Ross PJ, Maisey NR, Hughes S, Kwan W, Harari D. A comprehensive geriatric assessment screening questionnaire (CGA-GOLD) for older people undergoing treatment for cancer. Eur J Cancer Care (Engl). 2017 Sep;26(5). doi: 10.1111/ecc.12509. Epub 2016 May 1. PMID 27132979
- [Background] Parker SG, McCue P, Phelps K, McCleod A, Arora S, Nockels K, Kennedy S, Roberts H, Conroy S. What is Comprehensive Geriatric Assessment (CGA)? An umbrella review. Age Ageing. 2018 Jan 1;47(1):149-155. doi: 10.1093/ageing/afx166. PMID 29206906
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] McIsaac DI, Gill M, Boland L, Hutton B, Branje K, Shaw J, Grudzinski AL, Barone N, Gillis C; Prehabilitation Knowledge Network. Prehabilitation in adult patients undergoing surgery: an umbrella review of systematic reviews. Br J Anaesth. 2022 Feb;128(2):244-257. doi: 10.1016/j.bja.2021.11.014. Epub 2021 Dec 16. PMID 34922735
- [Background] Gillis C, Ljungqvist O, Carli F. Prehabilitation, enhanced recovery after surgery, or both? A narrative review. Br J Anaesth. 2022 Mar;128(3):434-448. doi: 10.1016/j.bja.2021.12.007. Epub 2022 Jan 7. PMID 35012741
- [Derived] Wang SK, Wang P, Wang W, Lu S. Multimodal prehabilitation combined with perioperative enhanced recovery after surgery care for older patients undergoing spinal fusion surgery in China: protocol for a multicentre randomised controlled trial (PRACTICE trial). BMJ Open. 2024 Dec 11;14(12):e088339. doi: 10.1136/bmjopen-2024-088339. PMID 39663170